CLINICAL TRIAL: NCT00000952
Title: A Phase I/II Study of Ritonavir Therapy in HIV-1 Infected Infants and Children
Brief Title: A Study of Ritonavir (an Anti-HIV Drug) in HIV-Positive Infants and Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 345; 10602 (Registry Identifier: DAIDS ES); PACTG 345
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Dose-Response Relationship, Drug; Drug Therapy, Combination; Zidovudine; HIV Protease Inhibitors; Ritonavir; Lamivudine; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Ritonavir
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
The study examines the safety and effectiveness of ritonavir (an anti-HIV drug), alone and in combination with other anti-HIV drugs, in HIV-positive children under 2 years of age. This study will also determine the most effective doses of ritonavir for future pediatric HIV studies.

Infants infected with HIV by their mothers experience faster disease progression than adults or older children. Treatment with anti-HIV drugs administered at an early age may slow disease progression in infant populations.

DETAILED DESCRIPTION:
As a group, vertically infected children experience more rapid disease progression than children infected at an older age or adults. The early administration of potent antiretroviral regimens might significantly impact the course of vertical HIV-1 infection.

Infants and children are stratified by age, representative of the developmental differences related to drug metabolism (Group I: at least 6 months - 2 years, Group II: 3-6 months, Group IIIA: 1 month - 10 weeks, IIIB: 1 month - less than 3 months). Within each age group there will be two possible dosage cohorts. All age groups will be enrolled simultaneously into dosage Cohort I, at the initial drug dosage. Progression to Cohort II (at a higher or lower drug dosage) will be decided according to safety, tolerance or viral load in Cohort I. All therapy for Group I/II, whether in Cohort I or II, will be introduced as follows: single dose of ritonavir on Day 0, ritonavir monotherapy through Day 7 AM and combination therapy from Day 7 PM through Week 104. All therapy for Group IIIA & IIIB, whether in Cohort I or II, will be introduced as follows: single dose of ritonavir on Day 0 AM and transition to combination therapy Day 0 PM through Week 104. NOTE: Progression to combination therapy for Group IIIA infants is dependent upon the results of the single-dose ritonavir pharmacokinetics (PK). If the patient is no longer at least presumed to be HIV-infected, he/she will be discontinued from the study. Replacement infants, who will not receive the single dose of ritonavir, will be acquired from Group IIIB infants; new infants that are either presumed HIV infected or have already been shown to be HIV-infected. Clinical evaluations are conducted and blood and urine samples collected regularly during the treatment period in order to quantify HIV-1 levels and determine body chemistries. Pharmacokinetic studies require additional blood sampling up to Week 16. [AS PER AMENDMENT 6/30/98: Pharmacokinetics data from Cohort I showed that the proposed Cohort II starting dose was too low. The dose for Cohort II is now increased. All subjects in Groups I, II, and III will begin combination therapy on Day 0 at the increased dose.] [AS PER AMENDMENT 3/13/00: The study has been extended for an additional 104 weeks, provided the patient's viral load is undetectable (below 400 copies/ml) at the end of the initial study period. While on the treatment extension, patients must continue their current schedule for study drug administration and completion of study visits.]

ELIGIBILITY:
Inclusion Criteria

Children may be eligible for this study if they:

* Are HIV-positive. (Infants under 3 months old presumed to be HIV-positive are eligible to participate in the single-dose phase of the study.)
* Are between the ages of 4 weeks and 2 years (consent of parent or guardian required).

Exclusion Criteria

Children will not be eligible for this study if they:

* Have an opportunistic (AIDS-related) infection within 2 months of study entry.
* Are allergic to 3TC and/or ZDV.
* Have received anti-HIV drugs for 6 to 12 weeks.
* Have any infections requiring treatment.
* Are experiencing wasting (significant weight loss).
* Have any malignancies (cancer).
* Have certain immune diseases, are being fed through a tube, or have HIV-related encephalopathy (a degenerative disease of the brain).

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60
Dates: Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ram Yogev, Study Chair; Ellen Chadwick, Study Chair
Locations (12):
- United States (12):
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Nyu Ny Nichd Crs, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Incarnation Children's Ctr., New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - St. Jude/UTHSC CRS, Memphis, Tennessee

REFERENCES:
- [Background] Scott ZA, Chadwick EG, Catalina MD, McManus M, Yogev R, Palumbo P, Britto P, Sullivan JL, Luzuriaga K. HIV-1-specific CD8+T cells in vertically infected infants: early responses and the effects of antiretroviral therapy. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 169)
- [Background] Zhao Y, Vetterick T, Lewis D, Yu M, Chadwick E, Yogev R, Coberly SK, Palumbo P. Genotypic mutations in the protease (Pr) and reverse transcriptase (RT) genes associated with antiretroviral resistance to combination therapy with ritonavir/AZT/3TC: a virological sub-study of PACTG 345. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 467)
- [Result] Chadwick EG, Rodman JH, Britto P, Powell C, Palumbo P, Luzuriaga K, Hughes M, Abrams EJ, Flynn PM, Borkowsky W, Yogev R; PACTG Protocol 345 Team. Ritonavir-based highly active antiretroviral therapy in human immunodeficiency virus type 1-infected infants younger than 24 months of age. Pediatr Infect Dis J. 2005 Sep;24(9):793-800. doi: 10.1097/01.inf.0000177281.93658.df. PMID 16148846